CLINICAL TRIAL: NCT00703963
Title: Improved Time in Therapeutic Range With Patient Self-Testing of Their INR Compared to Usual Care: A Randomized Controlled Trial
Brief Title: Improved Time in Therapeutic Range With Patient Self-Testing of Their INR Compared to Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Principal Investigator, Hartzell V. Schaff, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 07-001398
Record Dates: First submitted 2008-06-10; First posted 2008-06-24 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Management of Anticoagulation
Keywords: International normalized ratio (INR)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Subjects will be having their INR tested by their Primary Care Provider as often as their Care Provider dictates. This study phase is twelve weeks long beginning at the day of discharge from our hospital.
  Interventions: Other: Usual Care
- Patient Self Testing (Active Comparator): Subjects will be testing their INR at home using an FDA approved device (INRatio monitor by Hemosense) reporting their results to Quality Assured Services (QAS) via an 800 phone number; their Primary Care Provider will receive a fax with the INR result. We ask this group of patients to test at minimum one time a week, additional testing as requested by their Primary Care Provider. This phase lasts twelve weeks, beginning on the day of discharge from our hospital.
  Interventions: Device: INRatio monitor by Hemosense

INTERVENTIONS:
Device: INRatio monitor by Hemosense — Home testing monitor to test patients INR by placing a capillary drop of blood from the finger onto a test strip. The test strip is then inserted into the INRatio point-of-care self-testing coagulometer. After approximately 2 minutes of analysis, the INR value will be presented on the meter's display.
  Arms: Patient Self Testing
Other: Usual Care — Usual care is defined as that care currently received by patients into whom mechanical heart valves are placed. Typically, these patients undergo frequent checks of their INR level until the therapeutic range is achieved. Then periodic INR levels are drawn at the discretion of the managing physician.
  Arms: Usual Care

SUMMARY:
Patients who receive a mechanical heart valve to replace a diseased heart valve must take an anticoagulation medicine the rest of their lives, and monitor their level of anticoagulation. Until recently, the testing of the level of anticoagulation was performed at medical laboratories or hospitals.

The purpose of this study is to see if patients who test their level of anticoagulation by themselves at home and then call their doctor with the result have better control of their anticoagulation as compared to patients whose anticoagulation is checked only by their physician.

DETAILED DESCRIPTION:
Prosthetic replacement of diseased heart valves is a routine procedure, and mechanical heart valves have excellent hemodynamic performance and durability. However, mechanical valves are thrombogenic, necessitating lifelong anticoagulation. Hazards of anticoagulation include bleeding when it is excessive or thromboembolism when the intensity of anticoagulation is below the recommended level. Monitoring the level of anticoagulation is accomplished by analyzing the International Normalized Ratio. Until recently, this was performed at medical laboratories or hospitals, but recent literature suggests that patient self-testing of oral anticoagulation improves patient compliance, medical outcomes, and quality of life.

The objective of this study is to evaluate the time in therapeutic range of patients who self-test their INR compared to patients receiving the usual care. Additionally, we will evaluate the educational components and corollaries of self-testing.

Two hundred consecutively enrolled adults, having undergone implantation of a mechanical heart valve, will be randomized to either self-testing or usual care. Those randomized to the self-testing group will undergo self-testing instruction prior to hospital dismissal. For three months after hospital discharge, subject will record their INR results obtained by self-testing or as prescribed by their primary physician. They will then submit the record of the INR results and complete a survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received a mechanical valve while in our hospital
* Age > 18 years

Exclusion Criteria:

* Pregnant or lactating women
* Patients that have genetic clotting disorders such as Factor 5
* Physical disabilities (for example, poor eyesight, tremor, or other neurological disability) that would prevent the patient from being able to perform finger stick blood sampling. (Patients may not be excluded for physical disabilities if a care giver is willing to learn and assist with performing patient self-testing.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hartzell V Schaff, M.D. CS, Principal Investigator — Mayo Clinic
Locations (1):
- Saint Marys Hospital, Rochester, Minnesota, United States

REFERENCES:
- [Result] Thompson JL, Burkhart HM, Daly RC, Dearani JA, Joyce LD, Suri RM, Schaff HV. Anticoagulation early after mechanical valve replacement: improved management with patient self-testing. J Thorac Cardiovasc Surg. 2013 Sep;146(3):599-604. doi: 10.1016/j.jtcvs.2012.03.088. Epub 2012 Aug 24. PMID 22921821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic, Rochester, Minnesota from June 2007 to January 2009.
Period: Overall Study
Arm/Group | Usual Care | Patient Self Testing
Started | 100 | 100
Completed | 93 | 86
Not Completed | 7 | 14
Not completed — Withdrawal by Subject | 7 | 13
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Patient Self Testing | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Median (Full Range); unit: years] | 53 [19 to 84] | 55 [18 to 79] | 54 [18 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 33 | 73
  Male | 60 | 67 | 127
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Time in Therapeutic Range
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care | Patient Self Testing
Number analyzed (Participants) | 93 | 86
percentage of time | 48 (25) | 53 (27)
Statistical Analysis 1: Comparison: Usual Care vs Patient Self Testing; Statistical significance was defined as p < 0.05; Test type: Superiority or Other; p = 0.20, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Mean Percentage of INR Tests Within the Therapeutic Range
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: percentage of tests
Arm/Group | Usual Care | Patient Self Testing
Number analyzed (Participants) | 93 | 86
percentage of tests | 45 (22) | 52 (22)
Statistical Analysis 1: Comparison: Usual Care vs Patient Self Testing; Statistical significance was defined as p < 0.05; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mean Number of INR Tests Performed
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: INR tests
Arm/Group | Usual Care | Patient Self Testing
Number analyzed (Participants) | 93 | 86
INR tests | 10 (6) | 14 (9)
Statistical Analysis 1: Comparison: Usual Care vs Patient Self Testing; Statistical significance was defined as p < 0.05; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Subjects were followed up for 90 days after hospital dismissal.
Arm/Group | Usual Care | Patient Self Testing
Serious Adverse Events (participants affected / at risk) | 3/93 | 8/86
Other Adverse Events (participants affected / at risk) | 4/93 | 1/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=93) | Patient Self Testing (N=86)
Transient ischemic attack (Vascular disorders) | 1 | 2
Possible transient ischemic attack (Vascular disorders) | 1 | 0
Hemothorax (Vascular disorders) | 0 | 2
Evacuation of subdural hematoma (Vascular disorders) | 0 | 1
Bloody pericardial effusion (Vascular disorders) | 1 | 2
Pulmonary embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=93) | Patient Self Testing (N=86)
Temporary visual change (Eye disorders) | 2 | 0
Bleeding after shaving (Vascular disorders) | 1 | 0
Epistaxis (Vascular disorders) | 1 | 0
Bleeding scalp (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No